CLINICAL TRIAL: NCT01873703
Title: A Phase 2 Randomized Double-Blind Placebo-Controlled Study of Pracinostat in Combination With Azacitidine in Patients With Previously Untreated International Prognostic Scoring System (IPSS) Intermediate Risk-2 or High-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Phase 2 Study of Pracinostat With Azacitidine in Patients With Previously Untreated Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEI-003
Record Dates: First submitted 2013-05-22; First posted 2013-06-10 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Myelodysplastic Syndrome
Keywords: MDS; High risk myelodysplastic syndrome; Intermediate-2 Myelodysplastic syndrome; Untreated
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — SB939 compound; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pracinostat plus azacitadine (Experimental): 60 mg of pracinostat by mouth 3 times a week for 3 weeks followed by 1 week of rest repeated every 28 days.
  75 mg/m2 Azacitidine for 7 days of each 28 day cycle, via subcutaneous (SC) injection or intravenous infusion if SC injections are intolerable
  Interventions: Drug: pracinostat; Drug: Azacitidine
- Placebo with Azacitadine (Placebo Comparator): Placebo by mouth 3 times a week for 3 weeks followed by 1 week of rest repeated every 28 days.
  75 mg/m2 Azacitidine for 7 days of each 28 day cycle, via subcutaneous (SC) injection or intravenous infusion if SC injections are intolerable
  Interventions: Drug: Placebo; Drug: Azacitidine

INTERVENTIONS:
Drug: pracinostat — Histone deacetylase inhibitor (HDACi)
  Other Names: SB939
  Arms: pracinostat plus azacitadine
Drug: Placebo — Placebo
  Arms: Placebo with Azacitadine
Drug: Azacitidine — Active comparator 75 mg/m2 Azacitidine for 7 days of each 28 day cycle, via subcutaneous (SC) injection or intravenous infusion if SC injections are intolerable
  Other Names: Vidaza

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled study is to determine the safety and efficacy of pracinostat compared to placebo when combined with azacitidine, and FDA approved treatment for Myelodysplastic Syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Histologically or cytologically documented diagnosis of MDS (any French-American-British [FAB] classification subtype; that is classified as intermediate 2 (1.5 to 2.0 points) or high risk (≥2.5 points) according to the International Prognostic Scoring System risk category, with >5% and <30% blasts, and a peripheral blast count of <20,000
* Bone marrow aspirate smears and bone marrow biopsies within 28 days of first study treatment
* There must be a clinical indication for treatment with azacitidine.
* Previously untreated with hypomethylating agents (prior therapy with transfusions, hematopoietic growth factors, or immunosuppressive therapy is allowed)
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2
* Adequate organ function as evidenced by:

  1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x the upper limit of normal (ULN) (≤5 x ULN for patients with hepatic metastases
  2. Total bilirubin ≤1.5 x ULN or total bilirubin of 2, whichever is higher
  3. Serum creatinine <2 mg/dL, or creatinine clearance ≤1.5 x ULN
  4. QTcF interval ≤470 msec
* Female or male patients ≥18 years-of-age
* Male patients who are surgically sterile or willing to use adequate contraceptive measures or abstain from heterosexual intercourse during the entire study treatment period
* Female patients who are surgically sterile or post menopausal or female patients who are not of child-bearing potential and female patients of child-bearing potential who agree to use adequate contraceptive measures or abstain from intercourse during the study treatment period, who are not breastfeeding, and who have had a negative serum pregnancy test ≤7 days prior to first study treatment.
* Willingness and ability to comply with the trial and follow-up procedures

Exclusion Criteria:

* Received any of the following within the specified time frame prior to administration of study medication:

  1. Any investigational agent within 14 days or 5 half-lives prior to first study treatment, whichever is longer
  2. Previous therapy for malignancy within 21 days prior to first study treatment, including any chemotherapy, immunotherapy, biological or hormonal therapy (6 weeks for nitrosoureas or mitomycin C)
  3. Hydroxyurea within 48 hours prior to first study treatment
  4. Hematopoietic growth factors: erythropoietin, granulocyte colony stimulating factor (G-CSF), granulocyte macrophage colony stimulating factor (GM-CSF), or thrombopoietin receptor agonists at least 7 days (14 days for Aranesp) prior to study enrollment
  5. Major surgery within 4 weeks prior to first study treatment
* Patients that have not recovered from side effects of previous therapy
* Cardiopulmonary function exclusion:

  1. Current unstable arrhythmia requiring treatment
  2. History of symptomatic congestive heart failure (New York Heart Association Classes III or IV)
  3. History of myocardial infarction within 6 months of enrollment
  4. Current unstable angina
* Concomitant treatment with histone deacetylase (HDAC) inhibitors or drugs with significant action as HDAC inhibitors, such as valproic acid, is not permitted
* Clinical evidence of central nervous system involvement
* Patients with gastrointestinal (GI) tract disease, causing the inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis).
* Active infection with HIV or chronic hepatitis B or C
* Life-threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study
* Presence of a malignant disease within the last 12 months, with the exception of adequately treated in-situ carcinomas, basal or squamous cell carcinoma, or non-melanomatous skin cancer
* Inability (including psychological, familial, sociological, or geographical conditions) to comply with trial and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-06; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Estimate efficacy | 6 months
  Estimate the relative efficacy, measured by complete remission rate of treatment wiht pracinostat plus azacitidine versus placebo plus azacitidine

SECONDARY OUTCOMES:
Overall response rate | 6 months
  Estimate the overall response rate [ORR = CR + complete remission + partial response (PR)]
Hematologic Improvement | 6 months
  Estimate the overall hematologic improvement (HI) response rate by review of hematologic lab values each cycle including bone marrow blast counts, platelets and erythrocytes.
Duration of response | 6 months
  Estimate the duration of response
Progression free survival | 12 months
  Estimate the progression-free survival (PFS) duration of pracinostat plus azacitidine and the relative benefit of that combination versus placebo plus azacitidine as assessed by the PFS hazard ratio
Rate of leukemic transformation | 6 - 24 months
  Estimate the rate of leukemic transformation at landmark time points (6 months, 12 months, 18 months, and 24 months) using clinical review of hematologic lab counts each cycle
Overall survival | 6-24 months
  Estimate the overall survival (OS) duration of pracinostat plus azacitidine and the relative benefit of that combination versus placebo plus azacitidine as assessed by the OS hazard ratio
AE profile | 12 months
  Assess the adverse event (AE) profile of pracinostat and placebo when combined with azacitidine by clinical review of safety events by grade, relationship and event outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (24):
- United States (24):
  - Southern Cancer Center, Mobile, Alabama
  - Scripps Cancer Center, La Jolla, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Florida Cancer Specialist and Research Institute, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Indiana University Simon Cancer Ctr, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer at Johns Hopkins, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, Lansing, Michigan
  - Nebraska Methodist, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Weill Cornell Medical Center, New York, New York
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Cancer Center, Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Swedish Cancer Institute, Seattle, Washington

REFERENCES:
- See also: Sponsor website — http://MEIPharma.com